CLINICAL TRIAL: NCT07103369
Title: A Randomized, Double-Blind, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Preliminary Efficacy and Pharmacodynamics of SM17 in Chinese Healthy Subjects and Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Phase I Clinical Study to Evaluate SM17 in Chinese Healthy Subjects and Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SinoMab BioScience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM17-102; CTR20233129 (Other: Chinadrugtrials.org)
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Part 1: 3 single ascending dose (SAD) cohorts and 1 multiple dose (MD) cohort will be conducted sequentially, starting from the lowest dose SAD cohort, initiation of the following cohort will be upon judgement of safety review council(SRC) at least 7 days after the dosing of last cohort.
  Part 2: 2 doses of SM17 groups and placebo group will be enrolled and studied in parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- SAD cohort 1 (Experimental): single ascending dose cohort 1, participants(HVs) will receive 70mg of SM17 or placebo intravenously in this cohort with randomization ratio 6:2
  Interventions: Drug: SM17 for injection; Other: SM17 placebo for injection
- SAD cohort 2 (Experimental): single ascending dose cohort 2, participants(HVs) will receive 200mg of SM17 or placebo intravenously in this cohort with randomization ratio 6:2
  Interventions: Drug: SM17 for injection; Other: SM17 placebo for injection
- SAD cohort 3 (Experimental): single ascending dose cohort 3, participants(HVs) will receive 600mg of SM17 or placebo intravenously in this cohort with randomization ratio 6:2
  Interventions: Drug: SM17 for injection; Other: SM17 placebo for injection
- MD cohort (Experimental): multiple doses cohort, participants(HVs) will receive consecutive doses of 600mg of SM17 or placebo intravenously, once every 2 weeks in this cohort with randomization ratio 6:2
  Interventions: Drug: SM17 for injection; Other: SM17 placebo for injection
- SM17 lower dose group (Experimental): treatment group for participants (AD patients) to receive lower consecutive dose of SM17 （200mg）intravenously once every 2 weeks until end of treatment
  Interventions: Drug: SM17 for injection
- SM17 higher dose group (Experimental): treatment group for participants (AD patients) to receive higher consecutive dose of SM17 （200mg）intravenously once every 2 weeks until end of treatment
  Interventions: Drug: SM17 for injection
- placebo group (Placebo Comparator): control group for participants (AD patients) to receive placebo doses intravenously once every 2 weeks until end of treatment
  Interventions: Other: SM17 placebo for injection

INTERVENTIONS:
Drug: SM17 for injection — SM17 monoclonal antibody for intravenous infusion use
  Arms: MD cohort; SAD cohort 1; SAD cohort 2; SAD cohort 3; SM17 higher dose group; SM17 lower dose group
Other: SM17 placebo for injection — placebo to be compared with SM17, excipient solution of SM17 monoclonal antibody without protein
  Arms: MD cohort; SAD cohort 1; SAD cohort 2; SAD cohort 3; placebo group

SUMMARY:
This trial is a phase 1, randomized, double-blind, placebo-controlled trial conducted in Chinese Healthy Volunteers and Patients with moderate-to-severe Atopic Dermatitis

It aims to evaluate the safety, tolerability, pharmacokinetic characteristics and immunogenicity of single and multiple doses of SM17 injection in healthy subjects . It also aims to evaluate the safety, tolerability, pharmacokinetic characteristics, pharmacodynamic effect and immunogenicity as well as preliminary efficacy in AD patients.

DETAILED DESCRIPTION:
This trial consists of 2 parts:

Part 1 (Ph1a) trial of the study is a dose-ascending study to evaluate the safety, tolerability, pharmacokinetic characteristics of SM17 in Chinese healthy volunteers. Safety and PK profiles of SM17 in Chinese population will be established firstly in this study following single and multiple doses of SM17 injection, and possible differences to those of SM17 in US populations will also be evaluated.

Part2 (ph1b) trial of the study is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and preliminary efficacy of SM17 in treating patients with moderate-to-severe atopic dermatitis(AD) following multiple doses of SM17 injections at two doses level of SM17 or placebo. PK/PD profiles, immunogenicity profile of SM17 in AD patients will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers：

* Male or Female，19~55 years old
* BMI ≥18.5 and <28.0 kg/m² at the screening visit, with body weight ≥50 kg for males and ≥45 kg for females
* Non-smokers or former smokers who have quit for at least 6 months, with a smoking history of <10 pack-years for former smokers at the screening visit. No history of alcohol consumption or light alcohol consumption prior to the screening visit.
* No abnormalities or abnormalities of no clinical significance (NCS) in vital signs, physical examination, laboratory tests, or electrocardiogram (ECG) results during the screening period, QTcF <450 msec for male and QTcF <470 msec for female subjects.
* Use one medically approved contraceptive method during the trial and for 6 months after the trial ends (specific methods see Appendix 1); No plans to donate sperm/ova during the trial and for 6 months after the trial ends.
* informed consent.

Eligible patients must have a history of inadequate response or intolerance to treatment with topical AD medications.

* Male or female, 18 ~70 years old
* Atopic dermatitis (Hanifin & Rajka) at the screening visit with eczema symptoms reported over 1year
* Eczema Area and Severity Index (EASI) score ≥16 at the screening and baseline visits
* Investigator's Global Assessment (IGA) score ≥3 at the screening and baseline visits
* ≥10% body surface area (BSA) of AD involvement at the screening and baseline visits
* Baseline pruritus numerical rating scale (NRS) weekly average score ≥4
* Documented recent history (within 6 months before the screening visit) of inadequate response to topical AD medication(s) or for whom topical treatments are medically inadvisable (e.g. intolerance, because of important side effects, or safety risks)
* Have applied a stable dose of topical bland emollient (moisturizer) at least twice daily for at least 7 consecutive days immediately before randomization
* Willing and able to comply with all clinic visits and study-related procedures
* Able to understand and complete study-related questionnaires
* Signed written informed consent

Exclusion Criteria:

Healthy volunteers:

* Presence of psychiatric or legal incapacity, significant emotional problems at the screening visit, or anticipation of such issues during the study period.
* Regular alcohol consumption within 6 months prior to screening.
* History or evidence of any clinically significant medical condition, situation, or disease.
* Any laboratory parameter meeting the following criteria:

  1. Total bilirubin (TBIL) >1.5 × upper limit of normal (ULN)
  2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × ULN
  3. Serum creatinine (Cr) >1.5 × ULN
  4. White blood cell count below the lower limit of normal (LLN), deemed clinically significant and unsuitable for inclusion by the investigator at screening or baseline.
* History or current diagnosis of cardiovascular/cerebrovascular disease.
* Prior hospitalization for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection.
* Evidence of any active or suspected bacterial, viral, fungal, or parasitic infection within 4 weeks prior to screening. Subjects deemed at high risk for parasitic diseases are also excluded.
* Known diagnosis of Type I/II diabetes mellitus or prediabetes.
* Administration of live (attenuated) vaccines within 1 month prior to first dose.
* History of any malignancy within 5 years prior to screening (except successfully treated carcinoma in situ of the cervix or surgically excised non-melanoma skin cancer).
* Any known history of primary or secondary immunodeficiency disorders.
* Positive drug urine screen or alcohol consumption within 48 hours prior to screening.
* History or presence of hypersensitivity or idiosyncratic reactions to protein therapies, drugs, any component of SM17, or related compounds.
* Active infection including: Tuberculosis (TB), Hepatitis B, Hepatitis C, Human Immunodeficiency Virus.
* Use of any prescription or non-prescription medication within 14 days or 5 half-lives (whichever longer) prior to first SM17 dose.
* Tattoos, scars at/near the infusion site, or any other condition potentially interfering with infusion site examination, per investigator assessment.
* Blood/plasma donation (≥500 mL) or significant blood loss within 2 months prior to screening; planned donation during study. Bone marrow donation within 3 months prior to first dose.
* Inability to undergo protocol-required visits/procedures per investigator/subject knowledge.
* Current/recent participation in another investigational drug/device study.

AD patients:

* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study
* Laboratory abnormality for serum hemoglobulin, WBC, neutrophils, platelet, ALT/AST, TBIL, serum creatinine at screening or baseline
* HIV/HBV/HCV/TB positive
* ECG abnormality with clinical significance
* History of concomitant diseases: VKC/AKC, other skin diseases, active chronic or acute infection requiring treatment with systemic medications, malignancy within 5 yrs, other major diseases
* History of acute allergies, or known allergies to composition of monoclonal antibodies or excipients
* Treatments within 4 weeks before the baseline visit, or is likely to require such treatment(s) during the study treatment:
* systemic corticosteroids, Janus kinase inhibitors
* other immunosuppressive/immunomodulating drugs (cyclosporine, mycophenolate-mofetil, IFN-γ,, azathioprine, MTX..)
* traditional Chinese medicine
* Treatment with TCS, TCI, PDE-4 inhibitor, or other topical AD medications within 1 week before baseline
* New treatment of anti-histamine or ICS within 1 week before baseline ( stable doses of anti-histamine or ICS is allowed during study)
* Treatment with biologics, within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever is longer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent AEs in each cohort(Ph1a) | Day 0 to Day85 (SAD cohorts), Day 0 to Day 113 (MD cohort)
  Safety and tolerability of SM17 in Chinese healthy volunteers administrated with SM17 or placebo intravenously. Treatment emergent AE was any unfavorable or unintended medical occurrence in each subject, including any abnormal changes in vital signs or lab testing with clinical significance judged by investigators, that happened during the period of receiving or after receiving the investigational product.
Incidence of Treatment emergent AEs (TEAEs) in each treatment group(ph1b) | Week 0 to Week 16
  Safety and tolerability of SM17 in Chinese AD patients administrated with SM17 or placebo intravenously. Treatment emergent AE was any unfavorable or unintended medical occurrence in each subject, including any abnormal changes in vital signs or lab testing with clinical significance judged by investigators, that happened during the period of receiving or after receiving the investigational product. changes in vital signs and lab testing

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) in Chinese healthy volunteers | 12 weeks following SM17 dose （SAD） or last dose （MD）
  Serum Pharmacokinetic (PK) parameter of SM17 in Chinese healthy subjects administrated with SM17 intravenously
Immunogenicity | Baseline to 12 weeks following SM17/placebo dose (SAD) or last dose(MD)
  ADA positive rate in Chinese healthy volunteers
Area under the plasma concentration versus time curve (AUC) in Chinese AD patients | Week 0 (baseline) to Week 16
  Pharmacokinetic parameter obtained from Chinese patients with moderate-to-severe AD administrated with SM17 intravenously
Efficacy for treating AD - EASI50% | Week12, Week 16
  Portion of participants reaching response as EASI50(A 50% decrease in Eczema Area and Severity Index, which ranges from 0~72, and a deeper decrease means better outcome) in Chinese patients with moderate-to-severe AD administrated with SM17 intravenously
Efficacy for treating AD-EASI75% | Week12, Week 16
  Portion of participants reaching response as EASI75(A 75%50% decrease in Eczema Area and Severity Index, which ranged from 0~72, and a deeper decrease means better outcome) in Chinese patients with moderate-to-severe AD administrated with SM17 intravenously
Efficacy for treating AD-EASI90% | Week12, Week 16
  Portion of participants reaching response as EASI90(a 90% decrease in Eczema Area and Severity Index, which ranges from 0~72, and a deeper decrease means better outcome) in Chinese patients with moderate-to-severe AD administrated with SM17 intravenously
Efficacy for treating AD-EASI score change | Week2,4,6,8,10,12,16
  EASI(Eczema Area and Severity Index) score(ranges 0~72，higher score means worse disease condition) change from baseline and percentage change from baseline in Chinese patients with moderate-to-severe AD administrated with SM17 intravenously
Efficacy for treating AD-IGA 0/1% | Week12, Week16
  Portion of participants reaching response as IGA 0/1 in Chinese patients with moderate-to-severe AD administrated with SM17 intravenously. Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™） score ranges from 0 to 4, with lower scores indicating less severe AD. IGA 0/1 is defined as scores of 0 or 1, indicating a clear or almost clear AD presentation, and with at least 2-point reduction from baseline at time of assessment.
Efficacy for treating AD- PP-NRS | Baseline (Week0) to Week 16
  Change from baseline and Percentage change from baseline in PP-NRS weekly average score. PP-NRS is peak pruritus numeric rating scale, ranges 0~10, with higher score indicating a more severe itch condition. PP-NRS is assessed by patients to evaluate the peak pruritus condition for the past 24 hrs. A weekly average score is calculated as mean value of PP-NRS scores of 7 consecutive days prior to the point of assessments (need at least scores from 4/7 days available required to get a valid weekly average score).
Efficacy for treating AD-NRS-4% | Week2，4，6，8，10，12，16
  Portion of participants reaching response as NRS-4 in Chinese patients with moderate-to-severe AD administrated with SM17 intravenously. PP-NRS is peak pruritus numeric rating scale, ranges 0~10, with higher score indicating a more severe itch condition. NRS-4 is defined as at least 4 points reduction from baseline in weekly average score of PP-NRS. A weekly average score baseline is calculated as mean value of PP-NRS scores of 7 consecutive days prior to treatments (need at least scores from 4/7 days available to get a valid weekly average score baseline).
Efficacy for treating AD-BSA% | Week 2，4，6，8，10，12，16
  Change from baseline in Body Surface Area%（BSA%） with AD involvement, with a larger BSA% indicating a more severe disease condition.
Efficacy in treating AD-SCORAD | Week 4，8，10，12，16
  Change from baseline and percentage change from baseline in SCORAD (SCORing Atopic Dermatitis), ranges 0~103, with higher score indication a worse disease condition.
Efficacy for treating AD-POEM | Week2，4，6，8，10，12，16
  Change from baseline and Percentage change from baseline in POEM (Patient-Oriented Eczema Measure scores, range 0-28), with higher score indicating a worse disease condition.
Efficacy for treating AD-DLQI | Week2,4,6,8,10,12,16
  Change from baseline in DLQI score (Dermatology Life Quality Index, range 0~30, with higher score indicating a higher disease burden).
Immunogenicity | Week 0~16
  ADA positive rate in Chinese patients with moderate-to-severe AD treated by SM17/placebo intravenously

OTHER OUTCOMES:
PD biomarkers- total IgE | Week0, 4, 8, 10, 12, 16
  Serum total IgE concentration (mg/L) tested from Chinese patients with moderate-to-severe AD, treated by SM17/placebo
Peak Plasma Concentration (Cmax) in healthy volunteers and AD patients | 12 weeks following SM17 dose (SAD) or last dose( MD) for ph1a, 0~16 week for ph1b
  PK parameter(Cmax) obtained from Chinese Healthy volunteers and patients with moderate-to-severe AD administrated with SM17 intravenously
Time to peak (Tmax) | 12 weeks following SM17 dose (SAD) or last dose( MD) for ph1a, 0~16 week for ph1b
  PK parameter(Tmax) obtained from Chinese Healthy volunteers and patients with moderate-to-severe AD administrated with SM17 intravenously
Elimination half-life (T1/2) | 12 weeks following SM17 dose (SAD) or last dose( MD) for ph1a, 0~16 week for ph1b
  PK parameter(T 1/2) obtained from Chinese Healthy volunteers and patients with moderate-to-severe AD administrated with SM17 intravenously
Elimination Rate Constant (Kel) | 12 weeks following SM17 dose (SAD) or last dose( MD) for ph1a, 0~16 week for ph1b
  PK parameter(Kel) obtained from Chinese Healthy volunteers and patients with moderate-to-severe AD administrated with SM17 intravenously
Total drug clearance from plasma (CL) | 12 weeks following SM17 dose (SAD) or last dose( MD) for ph1a, 0~16 week for ph1b
  PK parameter(CL) obtained from Chinese Healthy volunteers and patients with moderate-to-severe AD administrated with SM17 intravenously
Apparent volume of distribution at steady state after extravascular administration (Vz) | 12 weeks following SM17 dose (SAD) or last dose( MD) for ph1a, 0~16 week for ph1b
  PK parameter(Vz) obtained from Chinese Healthy volunteers and patients with moderate-to-severe AD administrated with SM17 intravenously
PD biomarker- Eosinophil counts | Week0,2,4,6, 8, 10, 12, 16
  Serum Eosinophil counts tested from Chinese patients with moderate-to-severe AD, treated by SM17/placebo
PD biomarker- Tarc | Week0, 4, 8, 10, 12, 16
  Serum Tarc (CCL17) concentration (pg/mL) tested from Chinese patients with moderate-to-severe AD, treated by SM17/placebo
PD biomarker-Eotaxin-3 | Week0, 4, 8, 10, 12, 16
  Serum Eotaxin-3 (CCL-26) concentration (pg/mL) tested from Chinese patients with moderate-to-severe AD, treated by SM17/placebo
PD biomarker- Periostin | Week0, 4, 8, 10, 12, 16
  Serum Periostin concentration (ng/mL) tested from Chinese patients with moderate-to-severe AD, treated by SM17/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Xin-Hua Gao, MD, Principal Investigator — The First Hospital of China Medical University，Shenyang，Liaoning
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No